CLINICAL TRIAL: NCT06775561
Title: Precision Diagnosis and Therapy for Rare Diseases by Interpreting Non-coding Genomes (PARADIGM)
Brief Title: Precision Diagnosis and Therapy for Rare Diseases by Interpreting Non-coding Genomes
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PARADIGM; PNRR: M6/C2_CALL 2022 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Neuromuscular Diseases; Eye Diseases; Genetic Disease
MeSH Terms: conditions — Neuromuscular Diseases; Eye Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood and fibroblasts or muscle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genomic characterization of RGD patients with ED/NMD: * patients/relatives or parents of patients with a clinical diagnosis of rare eye and neuromuscular diseases
  * patients/relatives or parents of patients with inconclusive data from ESOMA and aCGH (no pathogenic/probable pathogenic variant) or detection of a single hit (a pathogenic or probable pathogenic variant) in an autosomal recessive gene from ESOMA (or aCGH) or no pathogenic or probable pathogenic variant but detection of a large region of genomic homozygosity surrounding a candidate gene
  * patients/relatives or parents of patients with detection of cryptic VUS (variants of uncertain significance) (splicing/regulatory/non-coding CNVs) in candidate genes or pathogenic cryptic variants in a selected number of representative cases.
  Interventions: Genetic: PARADIGM study aims to streamline the process from genomic characterization of RGD patients with ED/NMD to identification of the suitable personalized therapy.

INTERVENTIONS:
Genetic: PARADIGM study aims to streamline the process from genomic characterization of RGD patients with ED/NMD to identification of the suitable personalized therapy. — Samples are collected by UO1/UO2/UO3. DNA/RNA samples are sent to UO3 for genome and transcriptome sequencing. In vitro systems or patient-derived cell models are used for in vitro experimental validation (UO2) or development of therapeutical approaches (UO2/UO4). Samples of cases still undiagnosed after the combined sequencing and validation approaches undergo long-read sequencing by an outsourcing facility. Sequencing data are transferred to UO1 for bioinformatic analysis and may be deposited into RDconnect for still inconclusive cases. Variants of interest from bioinformatic analyses and in vitro validations are collectively discussed by UO1/UO2/UO3 to evaluate their clinico-molecular significance and to be selected for testing therapeutic approaches by UO2/UO4. Blue arrows and shapes denote samples and personal data, while green data that make no identifiable person.

SUMMARY:
PARADIGM study, funded by the PNRR research grant, will focus on Eye Diseases (ED) and Neuro-Muscular Diseases (NMD) as groups of genetically heterogeneous diseases which are extensively studied by the Partners partecipating in the project; indeed ED and NMD are well clinically and molecularly characterized and approachable by drug-testing options already assessed and implemented by PARADIGM partners. ED and NMD represent good and compatible disease models as:

* both are genetically heterogeneous disorders where missing heritability is likely to be hidden in non-coding variants;
* many of the individual genes accountable for the ED and NMD cause autosomal recessive forms, increasing the chance of finding regulatory/splicing variants

DETAILED DESCRIPTION:
UO1 (IRCCS Azienda Ospedaliero-Universitaria di Bologna, Coordinator) will coordinate the data collection and management protocols under fundamental ethical principles and relevant national, EU and international legislation; will set-up the bioinformatic data warehouse and deploy the workflows to analyze omics data analysis applying its own and published bioinformatic pipelines and will contribute to multi-omics data analysis.

UO2 (IRCCS Fondazione Istituto Neurologico Casimiro Mondino, Partner) will perform HiC/UMI-4C analyses and will contribute to the identification, validation and characterization of non-coding variants associated with RGDs, providing cellular and molecular genetic tools for the project to be tested in vitro or on patients' cell cultures from blood or skin. Only in specific cases (e.g. genes selectively expressed in the affected tissue), induced pluripotent stem cells (iPSCs) started from patients' fibroblasts will be used to generate 2D/3D cell models (e.g. retinal organoids) differentiated into the tissue of interes to dissect the molecular basis of unresolved RGDs.

UO3 (Azienda Ospedaliero-universitaria Luigi Vanvitelli, Partner) will carry out and integrate Genome Sequencing (GS) and transcriptome analysis on RNA from accessible tissues, e.g., cultured peripheral blood mononuclear cells (PBMCs), cultured fibroblasts (or fibroblast derived organoids), skeletal muscle (only when available in diagnostic routine).

UO4 (Università degli Studi di Napoli Federico II) will develop state-of-art gene therapy approaches to correct non-coding variants associated with RGDs, and test their efficiency in relevant retinal organoid models.

UO1, UO2, UO3 will be the clinical centers for recruitment of patients and collection of samples. This partnership gathers experts in the main omics, clinical geneticists, molecular biologists, and gene therapists, with massive experience in handling omics data, characterizing genetic variants for clinical purpose and developing therapeutics for genetic diseases up to the clinical stage.

ELIGIBILITY:
Inclusion Criteria:

* patients/relatives of patients with clinical diagnosis of NMD/ED;
* patients/relatives of patients with inconclusive ES and aCGH data (no pathogenic/likely pathogenic variant) or finding of only a single hit (a pathogenic or likely pathogenic variant) in an autosomal recessive gene by ES (or aCGH) or no pathogenic or likely pathogenic variant but detection of a large region of genomic homozygosity surrounding a candidate gene;
* patients/relatives of patients with a finding of cryptic VUS (splicing/regulatory/noncoding CNVs) in ED/NMD genes or pathogenic cryptic variants in a selected number of representative cases.
* Signed informed consent to participate in the study.

Exclusion Criteria:

- Trios or nuclear families where both unaffected parents do not consent to participate will be excluded (similarly, a minimum number of 3 affected family members will be needed in multigenerational pedigrees).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include:
  * patients previously in diagnostic routine, who have provided informed consent for storage and secondary use of their biological samples and for being recontacted; they will be informed about the current project and requested to provide a new specific informed consent;
  * patients' parents and/or other relatives (e.g. siblings, auncle/aunt);
  * age: from 0 years (newborns) with no upper age limit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Identification of genomic variants | 22 months
  To efficiently and reliably identify, and clinically interpret, cryptic genomic variants, representing the central challenge for the next decades of human genetics. The study will focus on ED and NMD conditions. The Diagnostic yield will be calculated as the proportion of the diagnosed cases over the total cases. Cases will be considered to be diagnosed when pathogenic or likely pathogenic genotype(s) will be identified and will be consistent with the patients clinical phenotype and segregation in the family.

SECONDARY OUTCOMES:
Evaluation of therapeutic efficiency | 24 months
  To develop and validate the preferred strategy for a treatment based on RNA therapeutics, CRISPR/Cas9-mediated genome editing or drug-repositioning. The therapeutic efficiency will be evaluated by transfection in HEK293 cells both at the DNA, RNA and protein level and the most efficient approach will be further side-by-side tested in 3D retinal organoids, in order to evaluate in more relevant models their ability to rescue the splicing defect as well as to ameliorate disease-specific morphological alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Pippucci, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No